CLINICAL TRIAL: NCT06668727
Title: Safety and Antiviral Activity of a Monoclonal Hepatitis B Antibody: a First-in-human Phase 1, Placebo-controlled, Single Dose Escalation Clinical Trial in Individuals with Chronic Hepatitis B Infection (The SAMBA Study)
Brief Title: Safety and Antiviral Activity of a Monoclonal Hepatitis B Antibody (The SAMBA Study)
Acronym: SAMBA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAMBA-001; 2023-508444-22 (EudraCT Number)
Record Dates: First submitted 2024-10-25; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis B
Keywords: Chronic hepatitis B; Experimental trial; Monoclonal antibodies
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Participants (n=4), will be enrolled in Group 1 (HepB mAb19 3 mg/kg or placebo, single dose) and randomized 3:1 to HepB mAb19 or placebo with each participant being dosed at least 72 hours apart. Following enrollment and administration of study drug in the first two participants, the Protocol Safety Review Team (PSRT) will review available safety data (including safety labs) and only following this review and in the absence of dose limiting toxicities (DLT), the remaining two participants in Group 1 will be enrolled and randomized to HepB mAb19 or placebo.
  Interventions: Drug: HepB mAb19
- Group 2 (Experimental): Participants (n=4), will be enrolled in Group 2 (HepB mAb19 10 mg/kg or placebo, single dose) and randomized 3:1 to HepB mAb19 or placebo with each participant being dosed at least 72 hours apart.
  Interventions: Drug: HepB mAb19
- Group 3 (Experimental): Participants (n=4), will be enrolled in Group 2 (HepB mAb19 30 mg/kg or placebo, single dose) and randomized 3:1 to HepB mAb19 or placebo with each participant being dosed at least 72 hours apart.
  Interventions: Drug: HepB mAb19
- Group 4 (Experimental): Participants (n=18) will enroll in Group 4 in an open-label fashion and will receive the MTD. Enrollment in Group 4 will begin after all 4 participants enrolled in the preceding dose group reach at least 28 days, none of the dose escalating halting criteria outlined above occur, and following review of available safety data by the PSRT
  Interventions: Drug: HepB mAb19

INTERVENTIONS:
Drug: HepB mAb19 — The study has two parts:
  Part A will involve administering a single ascending dose of HepB mAb19 or placebo using a randomized, double-blind method in Groups 1-3 at dose levels of 3, 10, and 30 mg/kg. Participants enrolled in Groups 1-3 will be randomized at a 3:1 ratio to receive HepB mAb19 or placebo. Part B will assess the maximum tolerated dose (MTD) in Group 4 in an openlabel fashion. Participants will receive HepB mAb19 at MTD.

SUMMARY:
Hepatitis B virus (HBV) remains a major global health problem with an estimated 257 million people living with the infection worldwide. Chronic HBV (CHB) is a major cause of liver cirrhosis and hepatocellular carcinoma. While antiviral therapies are available and suppress viral levels, treatment is long-term, does not clear the infection and rarely leads to long-term control once discontinued. Moreover, treatment access is not ideal on a global level with less than 10% of people in need receiving treatment. Although a strategy that eliminates all viral particles from the body represents the "holy grail" of HBV therapy, a strategy that leads to HBsAg loss and allows patients to stop treatment is highly desirable. New strategies to achieve either complete viral clearance or a state of viral control without the need for long-term treatment are being developed, including approaches to restore immune responses. Antibodies are key modulators of immune responses because of their dual functionality. In addition to directly targeting a viral antigen, antibodies differ from direct antivirals in that they can recruit other immune cells to eliminate infected cells and accelerate viral clearance.

This study will evaluate the safety and pharmacokinetics of a monoclonal antibody that was isolated from an HBV-vaccinated individual, HepB mAb19, as well as its potential effects on viral levels and antiviral immune responses in individuals living with CHB.

DETAILED DESCRIPTION:
Along with persistence of viral antigens, impaired HBV-specific immunity contributes to chronicity of infection. Chronic HBV (CHB) is characterized by depletion or functional impairment of HBV-specific T cells, resulting in defective proliferation and cytokine production, as well as impaired production of antibodies against HBsAg, with an expansion of atypical memory B cells. The importance of host immunity for HBV clearance is well recognized, but the critical immunological events required to achieve functional cure are not fully understood. Persistent high HBsAg levels along with dysfunctional immunity has raised the possibility that HBsAg itself is immunoregulatory in HBV infection. Chronic exposure to high levels of HBsAg may render HBV-specific T cells overly activated and functionally tolerated. Thus, decreasing serum HBsAg could be a valuable therapeutic strategy, due to its potential to alleviate functional exhaustion and confer immune control.

In parallel, antibodies to HBsAg are associated with successful vaccination and recovery from acute infection. Indeed, a difference between chronically infected and naturally recovered individuals is a robust polyclonal B cell response to HBsAg. Whether these associations reflect an etiologic role for anti-HBV neutralizing antibodies is not known. However, depletion of antibody producing B lymphocytes in CHB patients by rituximab is associated with HBV reactivation, indicating that B cells or their antibody products are playing a significant role in controlling the infection. The only immunomodulatory therapy currently available to treat CHB, IFN-α, is effective in only 30% of people, with marked differences observed across HBV genotypes being most effective against HBV genotype A and B infections.New therapeutic strategies that interfere with viral persistence and ongoing immune dysregulation with the goal to achieve a functional cure are needed. Several strategies are in clinical development including antiviral (e.g.small interfering RNA) (siRNA) and nucleic acid polymers (NAPs), and immune restoration approaches (e.g. therapeutic vaccination, toll-like receptor agonists, checkpoint blockade inhibitors and passive immunotherapy with anti-HBs antibodies).

Antibodies are among the key modulators of immunity and are uniquely attractive pharmaceutical agents because of their dual functionality. In addition to targeting a specific epitope with their variable domains, antibodies differ from direct antivirals in that they can recruit immune effector functions through their Fc domains. In addition to accelerating clearance of viruses andinfected cells through phagocytosis or direct cellular cytotoxicity, antigen-antibody immune complexes are also potent immunogens that can foster development of host immune responses. For example, antibody-based cancer therapies eliminate malignant cells and induce adaptive T cell immunity, and have dramatically increased the number of individuals that control and survive malignant diseases. Whether the same concepts are applicable to the management of chronic viral infections is an area of active investigation, particularly in the HIV-1 field.

In CHB, antibodies have the potential to enhance clearance of HBsAg. Although studies in transgenic animals indicate that T cell tolerance to HBsAg is durable and difficult to reverse, the models are not entirely reflective of human infection.

Whether antibody therapy can restore some aspects of HBV-specific T cell immunity in humans has not been determined. Immunotherapy with HBsAg-specific antibodies has shown some direct HBsAg suppression effects in clinical studies. However, the HBsAg antibodies that were evaluated only led to short term decline in HBsAg levels in CHB patients, that were very similar to the effects of treatments based on hepatitis B immune globulin (HBIG). More potent antibodies with long-lasting effects on circulating HBsAg and potential to modulate and restore HBV-specific immune responses are needed to evaluate the role of immunotherapy in CHB treatment and remission.

This study aims to evaluate the safety, maximal tolerated dose, pharmacokinetics (PK) and antiviral effects of a highly potent neutralizing human monoclonal antibody (mAb), HepB mAb19, that targets HBV S-protein in individuals with CHB. Safety, PK and virologic data generated by this study will guide the selection of a dosing regimen for subsequent multidose studies in individuals with CHB, in combination with standard HBV antiviral therapy and/or other investigational products, including other anti-HBs mAbs.

HepB mAb19 is a human mAb of Immunoglobulin G (IgG) 1kappa isotype that specifically binds to the "a" determinant of the extracellular loop of the HBV surface antigen (HBsAg). HepB mAb-19 was isolated and cloned from an HBsAg vaccinated individual at the Rockefeller University. The naturally occurring antibody was modified by two one-amino acid substitutions. These substitutions enhance the antibody binding affinity to the neonatal Fc receptor, prolonging its half-life in vivo, but do not interfere with antigen binding or with affinity to Fc gamma receptors.

To assess the efficacy of anti-HBV antibodies in vivo, researchers used human liver chimeric FNRG mice, which can sustain HBV infection. They tested two antibodies, HepB mAb20 and HepB mAb07, as pre-exposure prophylaxis. Both antibodies successfully prevented HBV infection in these mice, while all control mice became infected. In mice with established HBV infections, HepB mAb20, HepB mAb07, and HepB mAb19 stabilized viremia but did not eliminate it entirely. Over time, some mice treated with mAb20 and mAb07 developed an increase in viremia, attributed to the emergence of the G145R escape mutation. Notably, HepB mAb19 did not lead to such escape mutations, suggesting higher resistance.

Further, combination therapies targeting different viral epitopes were evaluated. While a HepB mAb06 + HepB mAb07 combination showed partial resistance to escape mutations, it still allowed the emergence of mutations. In contrast, combinations such as HepB mAb17 + HepB mAb19 and a triple therapy (HepB mAb16, HepB mAb17, HepB mAb19) successfully controlled viremia and prevented escape mutations. These findings indicate that monotherapy may lead to escape mutations, while well-chosen antibody combinations can improve viral control, potentially enhancing immune response during antiviral therapy

A GLP-compliant study on HepB mAb19 tested cross-reactivity in normal human and rat tissues, revealing limited cytoplasmic binding in specific cells, mainly in acinar epithelial cells in human salivary glands and various rat tissues. Since the binding was cytoplasmic, it is unlikely to have toxicological significance. A 25-day toxicology study in rats (doses 0, 4, 15, or 60 mg/kg IV) showed no adverse effects or significant changes in clinical or lab parameters, establishing the no-observed-adverse-effect-level (NOAEL) at 60 mg/kg. HepB mAb19 showed dose-proportional peak concentration and stable half-life of 13-16 days, with a 4-fold exposure increase upon repeated dosing.

Our hypothesis is that intravenous administration of HepB mAb19 during suppressive nucleos(t)ide therapy will be safe and well tolerated, will lead to decreased levels of circulating HBsAg, and enhance host innate and adaptive immune responses to HBV.

The study has two parts:

Part A: In part A, a single dose of HepB mAb19 or placebo is administered by randomization into three different dose groups. Gradually higher doses of HepB mAb19 will be used, meaning that participants in group 1 will receive a low dose (3 mg/kg), which will be assessed for safety before a single dose of 10 mg/kg and 30 mg/kg are tested under the same principle. Participants in each group 1-3 will be randomized in a 3:1 ratio to receive either HepB mAb19 or placebo (normal saline).

Part B: Based on part A, the maximum tolerated dose (MTD) of HepB mAb19 will be established. This dose will subsequently be used in part B, where a fourth group of 18 individuals will receive HepB mAb19 without randomization.

Participants will undergo safety assessments 1, 3, and 7 days after the administration of the trial antibody or placebo infusion, then weekly through to week 4, and finally at weeks 8, 12, 24, 36, and 48.

Blood samples will be collected during study visits. These blood samples will be used for analyses of safety, how HepB mAb19 is absorbed in the body, the effects of HepB mAb19 on HBV, and the immune system's response to it. Blood samples will be collected on day 0 before the administration of HepB mAb19, at the end of the antibody or placebo infusion, after 1, 3, and 7 days, and during subsequent follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 to ≤ 70;
* HBV infection confirmed by positive HBsAg for ≥6 months;
* On HBV-active nucleos(t)ide therapy for ≥6 months without change in NRTI in the previous 3 months;
* The following laboratory values 49 days prior to study entry (day 0):
* HBV DNA below lower limit of quantification;
* HBs antibody negative;
* HBeAg negative;
* Ability and willingness to provide informed consent.
* For participants who can become pregnant (i.e., participants who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy), negative serum or urine pregnancy test at screening and on day 0 (study entry).
* Participants who can become pregnant must agree to use two methods of contraception, one of which must be from the highly effective methods for contraception listed below. Barrier methods of contraception are permitted for the second method of contraception. Contraception must be used from 10 days prior to study entry and during study follow up. Acceptable methods of contraception include:
* Contraceptive subdermal implant;
* Intrauterine device or intrauterine system;
* Combined estrogen and progestogen oral contraceptive;
* Injectable progestogen;
* Contraceptive vaginal ring;
* Percutaneous contraceptive patches;
* Partner sterilization with documentation of azoospermia prior to the participant's entry into the study, and this partner is the sole partner for that participant. The documentation of partner sterility can come from the site personnel's review of medical records or medical history interview provided by the participant or the partner. Self-reported documentation of reproductive potential should be entered in the source documents.
* Participants who can impregnate a partner and who are engaging in sexual activity that could lead to pregnancy must agree to use condoms from 10 days prior to study entry and during study follow up to avoid impregnating a partner who can get pregnant.

Exclusion Criteria:

* Clinical symptoms, imaging studies or liver histology suggestive of advanced fibrosis (exclude fibrosis grade 3 and 4 by FibroScan) (Fibroscan®< 9 kpa) 12 months prior to entry or done at the pre-infusion visit. Note: If FibroScan results are not available, imaging will be performed at the preinfusion visit.
* Presence of a LI-RADS4 or 5 liver lesion on imaging 12 months prior to entry or done at pre-infusion visit, if prior results not available.
* Alpha fetoprotein >20 ng/ml. Note: Alpha-fetoprotein (AFP) above normal but < 20 is acceptable for entry if earlier AFP levels (older than 6 months) are within normal range and imaging is negative in last 3 months).
* HIV-1, HCV or hepatitis delta virus infection 12 months prior to entry or done at screen, if prior results not available;
* History of hematopoietic stem cell transplant or solid organ transplant;
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, monoclonal antibody or vaccine, or multiple drug allergies (non-active hay fever is acceptable);
* History of cardiovascular disease (e.g., cardiac insufficiency, coronary artery disease, cardiomyopathy, congestive heart failure, family history of congenital long QT syndrome, family history of sudden death);
* History or presence of clinically significant Electrocardiogram (ECG) abnormalities based on the average of the triplicate ECG recordings (e.g., PR interval >210 ms, QT corrected for heart rate using the Fridericia's correction factor [QTcF] > 450 ms for males and QTcF >470 ms for females);
* History of systemic corticosteroids, immunosuppressive anti-cancer, systemic interferons or interleukins 6 months prior to entry;
* History of chronic liver disease from another cause, ICD, or autoimmune diseases that in the opinion of the investigator would preclude participation;
* Any significant acute infection (e.g. influenza, COVID-19) or any other clinically significant illness 2 weeks prior to entry.
* Laboratory abnormalities in the parameters listed below:
* Absolute neutrophil count <1,000 /mm3
* Hemoglobin <10 gm/dL (6.21 mmol/L)
* Platelet count <150,000 /mm3
* ALT >2.0 x Upper normal limit (ULN)
* AST >2.0 x ULN
* Total bilirubin >1.5 ULN (except individuals with known Gilbert's)
* Albumin <3.5 gm/dL
* Estimated glomerular filtration rate (eGFR) <70 mL/min
* INR ≥1.2
* Pregnancy or lactation;
* Any vaccination 2 weeks prior to entry;
* Receipt of anti-HBV mAb therapy of any kind in the past (including HBIG);
* Participation in another clinical study of an investigational product currently or 12 weeks prior to, or expected participation during this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2027-08-26 (Estimated); Study Completion 2027-08-26 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From enrollment to the end of follow up at 48 weeks
  Safety and tolerability evaluation will be done by recording of adverse events. The DAIDS AE Grading Table Corrected version 2.1 (July 2017) will be used to grade adverse events. In addition, the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grading scale will be used for reporting and grading adverse events related to infusion reactions and cytokine release syndromes within 24 hours of the start of IP or placebo administration that are considered administration reactions or cytokine release syndromes.
Pharmacokinetic profile | From enrollment to the end of follow up at 48 weeks
  HepB mAb19 levels in serum will be measured by a validated sandwich ELISA method developed and performed by Celldex Therapeutics. HepB mAb19 levels will be measured before and at the end of the administration, at 3 and 6 hours, 1, 3, 7 days and on weeks 2, 3, 4 weeks after administration, and at later time points during follow up.
Pharmacokinetic profile | From enrollment to follow up at 48 weeks
  Assesment of HepB mAb19 elimination half-life (t1/2)
Pharmacokinetic profile | From enrollment to follow up at 48 weeks
  Assesment of clearance (CL/F) of HepB mAb19
Pharmacokinetic profile | From enrollment to follow up at 48 weeks
  Calculation of volume of distribution (Vz/F)
Pharmacokinetic profile | From enrollment to follow up at 48 weeks
  Calculation of area under the curve (AUC) for HepB mAb19
Pharmacokinetic profile | From enrollment to follow up at 48 weeks
  Calculation of HepB mAb19 decay curve
Maximum tolerated dose | From enrollment to follow up at 48 weeks
  To establish the maximum tolerated dose (MDT)

SECONDARY OUTCOMES:
HBsAg levels | From enrollment to the end of follow up at 48 weeks
  To determine the effects of HepB mAb19 on serum HBsAg levels
HepB mAb19 antibodies | From enrollment to the end of follow up at 48 weeks
  To assess the frequency induced anti-HepB mAb19 antibodies

OTHER OUTCOMES:
HBV markers | From enrollment to the end of follow up at 48 weeks
  To evaluate effects on other HBV markers such as HBV DNA, HBV RNA and HBcore-related Ag (HBcrAg)
HbsAg and HbeAg seroconversion | From enrollment to the end of follow up at 48 weeks
  To evaluate the frequency of HBsAg and HBeAg seroconversion following HepB mAb19 administration
HBV specific immune responses | From enrollment to the end of follow up at 48 weeks
  To evaluate HBV-specific T and B cell immune responses following administration of HepB mAb19.
Innate immune responses | From enrollment to the end of follow up at 48 weeks
  To evaluate innate immune responses following administration of HepB mAb19
Inflammatory markers | From enrollment to the end of follow up at 48 weeks
  To evaluate effects on inflammatory markers, such as soluble CD14, IL-6, Creactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Ole S. Søgaard, MD, Professor, Principal Investigator — Infectious Diseases, Aarhus University Hospital, Denmark
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No